CLINICAL TRIAL: NCT04584762
Title: Automated Variable Pattern Insufflator Device (AVPI) for the Acute Treatment of Migraine: a Prospective, Randomized, Double-blind, Parallel Group, Sham-controlled Clinical Trial
Brief Title: Automated Variable Pattern Insufflator Device (AVPI) for the Acute Treatment of Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nocira, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NC05
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, parallel group, sham-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Sham treatment (Sham Comparator): The AVPI device software is set in "sham mode" which does not deliver the therapy to the subject. Neither the subject or the investigator is aware of which mode is being used.
  Interventions: Device: Automated Variable Pressure Insufflation
- Active Treatment (Experimental): The AVPI device software is set in "active mode" which delivers the therapy to the subject. Neither the subject or the investigator is aware of which mode is being used.
  Interventions: Device: Automated Variable Pressure Insufflation

INTERVENTIONS:
Device: Automated Variable Pressure Insufflation — Acute migraine treatment

SUMMARY:
Randomized, sham-controlled, double-blind study for acute migraine attacks. Randomized to active treatment and sham treatment arms for the first treatment. Optional second active treatment. Follow up at 0, 2 and 24 hours post-treatment.

DETAILED DESCRIPTION:
Randomized, sham-controlled, double-blind study for acute migraine attacks.

Treatment Phase:

• ≤60 days to present at clinic for treating up to 2 migraines (at least 48 hours apart). First treatment is randomized between active treatment and sham treatment. Second optional treatment is open-label.

Post-Treatment Follow-up Phase:

* 24 hours after initiating treatment, for each of up to two migraine treatments, for conducting post-treatment follow-up assessments of migraine symptoms.
* 30, 60, and 90 days following the first migraine treatment for migraine diary assessments (and MIDAS assessment at 90 days)

Collection of migraine diaries at 30, 60, & 90 days post enrollment. Collection of MIDAS data at 60 and 90 days post treatment.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at the time of the baseline visit.
2. Episodic migraine with or without aura diagnosed according to the International Classification of Headache Disorders 3 beta diagnostic criteria.
3. Migraine onset before the age of 50 years
4. Migraine present for at least 1 year at the time of the Baseline Visit.
5. Frequency of 1-12 migraine attacks per month in each of the 2 months prior to screening.
6. Willingness, ability, and commitment to participate in baseline and follow-up evaluations without concurrent participation in another clinical trial.
7. Signed patient informed consent form.

Exclusion Criteria:

1. Prior or current diagnosis of migraine with brainstem aura, hemiplegic migraine, retinal migraine, migraine aura without headache, vestibular migraine.
2. Use of acute headache medication within previous 48 hours of treatment visit (for each treatment visit).
3. Use of acute medication for headache on >15 days per month in the 3 months prior to the Baseline Visit.
4. Change in migraine preventive therapies or dosage within the preceding 1 month of Baseline Visit.
5. Use of an opioid or barbiturate on more than 4 days per month in each of the 3 months prior to the Baseline Visit.
6. Other primary headache disorder, other than tension-type headache on 3 or fewer days per month.
7. History of secondary non-migraine headache disorders.
8. Medical history of Meniere's disease; endolymphatic hydrops; loss of hearing in either ear that is either complete, requires a hearing aid, or has deteriorated noticeably over the past year; ear surgery (including ear tubes); chronic continuous or current tinnitus; superior canal dehiscence.
9. Discomfort, infection, or other abnormal symptoms or disorders of either ear within 1 month prior to the enrollment Screening or Treatment Visit.
10. Pregnant or trying to become pregnant.
11. Unable to provide informed consent.
12. Inability to present to the medical clinic for study treatment during a migraine attack.
13. Unable or unlikely to follow instructions for proper use of the device.
14. Presence of any condition or state that would prevent the subject from sitting or lying down during the course of the treatment (up to 30 minutes).
15. History of receiving ear pressure therapy (insufflation) to treat any condition.
16. Personal or family affiliation as a service provider (e.g. employee, contractor, consultant, or volunteer) with a migraine treatment device company other than the study sponsor.
17. Perforated or compromised tympanic membrane, and which is confirmed by otoscope inspection by the Investigator before or upon presentation of the subject for the Treatment Visit.
18. Any other information about the subject's medical condition that, in the reasonable professional judgement of the Investigator, may adversely affect the intended safety or results of the treatment as intended and as a reasonable basis to exclude the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Pain Freedom Rates - active | 2 Hours post treatment
  Pain freedom rates (PFR)

CONTACTS AND LOCATIONS:
Overall Officials: David George, Study Director — Nocira, LLC
Locations (3):
- United States (3):
  - Regen Pain and Wellness, Scottsdale, Arizona
  - Murray Chiropractic Neurology, St. Petersburg, Florida
  - StudyMetrix, Saint Charles, Missouri

IPD SHARING:
Plan to Share IPD: No